CLINICAL TRIAL: NCT04059406
Title: A Phase 2a, Randomized, Open-Label Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ISIS 702843 Administered Subcutaneously to Patients With Non-Transfusion Dependent β-Thalassemia Intermedia
Brief Title: Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Sapablursen (Formerly ISIS 702843, IONIS-TMPRSS6-LRx)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Favorable safety and tolerability were seen, but efficacy results in the mid-stage study did not meet Ionis' minimum target product profile to justify further development.
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 702843-CS2; 2019-003505-96 (EudraCT Number)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Beta Thalassemia Intermedia
Keywords: Thalassaemia; Beta Thalassemia; IONIS TMPRSS6-LRx
MeSH Terms: conditions — beta-Thalassemia; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort A: Sapablursen (Experimental): Subjects initially received 30 mg/0.3 mL of sapablursen by (subcutaneous) SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg once every 4 weeks.
  Interventions: Drug: sapablursen
- Cohort B: Sapablursen (Experimental): Subjects initially received 50 mg/0.5 mL of sapablursen by SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg once every 4 weeks
  Interventions: Drug: sapablursen
- Cohort C: Sapablursen (Experimental): Subjects initially received 80 mg/0.8 mL of sapablursen by SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg once every 4 weeks.
  Interventions: Drug: sapablursen

INTERVENTIONS:
Drug: sapablursen — sapablursen administered subcutaneously
  Other Names: ISIS 702843; IONIS TMPRSS6-LRx

SUMMARY:
The purpose was to evaluate the efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics of sapablursen administered subcutaneously to participants with non-transfusion dependent β-Thalassemia Intermedia.

DETAILED DESCRIPTION:
This was a multi-center, randomized, open-label study in up to 29 participants. The duration of participation for each subject in the study was approximately 29 months and included an approximately 2-month screening period, a 24-month treatment period, and a 3-month post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with study procedures
* Clinical diagnosis of Beta-Thalassemia Intermedia with genotypic confirmation
* Non-transfusion dependent, as defined by: no more than 6 transfusions in the past 12-month period, and no transfusions in the 8-week period prior to Day 1
* Mean Hb within the range of 6.0-10.0 g/dL, inclusive at Screening
* LIC within the range of 3.0-20.0 mg Fe/g dry weight, inclusive
* If using chelators, must be on a stable dose for at least 3 months with liver iron concentration (LIC) > 5.0 mg iron (Fe) per gram of dry weight of liver (Fe/g) dry weight and serum ferritin > 300 nanograms per milliliter (ng/mL)
* Females must be non-pregnant and non-lactating, and either surgically sterile or postmenopausal
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method

Exclusion Criteria:

* Clinically significant abnormalities in lab values, medical history, or physical examination
* α-globin gene triplication
* Symptomatic splenomegaly
* Platelet count < lower limit of normal (LLN) or > 1,000 x 10^9/L
* Significant concurrent/recent coagulopathy, history of non-traumatic significant bleeding; history of immune thrombocytopenic purpura (ITP); current use of SC anti-coagulants; history of thrombotic events, including stroke or DVT
* Clinically significant renal, liver or cardiac dysfunction
* Uncontrolled hypertension (> 140 mm Hg systolic or > 90 mm Hg diastolic)
* Fasting blood glucose > 2.0 × upper limit of normal (ULN)
* Inability to have a magnetic resonance imaging (MRI) scan
* Known history or positive test for human immunodeficiency virus (HIV), hepatitis C (HCV), or hepatitis B (HBV)
* Active infection requiring systemic antiviral or antimicrobial therapy
* Regular excessive use of alcohol
* Recent start of hydroxyurea (6 months prior to Day 1)
* Treatment with or recent exposure to another investigational drug, biological agent, antisense oligonucleotide (ASO), small interfering ribonucleic acid (siRNA), or device within 1 month of Screening, or 5 half-lives of investigational agent, whichever is longer; or treatment with or exposure to:

  * sotatercept (ACE-011), luspatercept (ACE-536), or ruxolitinib within 4 months of Screening
  * hematopoietic stimulating agents or any hypoxia-inducible factor prolyl hydroxylase inhibitors within 8 weeks of Day 1
  * prior bone marrow transplant, stem cell transplant, or gene therapy
* Surgery associated with significant blood loss within 4 months of Screening, splenectomy within 12 months of Screening, or splenectomy scheduled during treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Greece (3):
  - Aghia Sophia General Children's Hospital, Athens, Attica
  - University General Hospital of Patras, Patra, Peloponnese
  - Koutlimbaneio & Triantafylleio General Hospital of Larissa, Larissa, Thessaly
- Chronic Care Center, Hazmiyeh, Lebanon
- Thailand (7):
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - King Chulalongkorn Memorial Hospital, Pathum Wan
  - Naresuan University Hospital, Phitsanulok
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (5):
  - Cukurova Üniversitesi Tıp Fakültesi, Adana
  - Hacettepe Üniversitesi Tıp Fakültesi, Ankara
  - Akdeniz University Faculty of Medicine, Antalya
  - Ege Universitesi Tip Fakultesi, Izmir
  - İstanbul Üniversitesi - Istanbul Tıp Fakültesi, Topkapı

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 15 investigative sites in Australia, Greece, Lebanon, Thailand, and Turkey from 24 September 2020 to 28 March 2023.
Pre-assignment Details: A total of 71 participants were screened with a diagnosis of β-Thalassemia, of which 29 participants were enrolled in either cohorts A, B, or C to receive sapablursen.
Groups:
- Cohort A: Sapablursen: Subjects initially received 30 mg/0.3 mL of sapablursen by SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg.
- Cohort B: Sapablursen: Subjects initially received 50 mg/0.5 mL of sapablursen by SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg.
- Cohort C: Sapablursen: Subjects initially received 80 mg/0.8 mL of sapablursen by SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg.
Period: Overall Study
Arm/Group | Cohort A: Sapablursen | Cohort B: Sapablursen | Cohort C: Sapablursen
Started | 6 | 6 | 17
Completed | 1 | 1 | 2
Not Completed | 5 | 5 | 15
Not completed — Early Treatment Termination | 5 | 5 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Sapablursen | Cohort B: Sapablursen | Cohort C: Sapablursen | Total
Number analyzed (Participants) | 6 | 6 | 17 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (12.12) | 31.7 (10.44) | 32.0 (10.88) | 32.6 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 10 | 18
  Male | 2 | 2 | 7 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 5 | 9 | 17
  Race: Asian | 3 | 1 | 8 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 6 | 6 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a ≥1.0 Grams Per Deciliter (g/dL) Increase From Baseline in Hemoglobin (Hb) at Week 27
Description: Blood hemoglobin
Time Frame: Baseline and Week 27
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of sapablursen and who had at least 1 Hb assessment collected after Day 1. Here, the "overall number of participants analyzed" signifies the number of participants available for analysis for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Sapablursen | Cohort B: Sapablursen | Cohort C: Sapablursen
Number analyzed (Participants) | 6 | 6 | 15
percentage of participants | 0 [0.0 to 45.9] | 0 [0.0 to 45.9] | 6.7 [0.2 to 31.9]

2. Secondary Outcome: Percentage of Participants With a ≥1.5 g/dL Increase From Baseline in Hb at Week 53
Description: Blood hemoglobin
Time Frame: Week 53
Population: FAS included all randomized participants who received at least 1 dose of sapablursen and who had at least 1 Hb assessment collected after Day 1. Here, the "overall number of participants analyzed" signifies the number of participants available for analysis for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A: Sapablursen: Subjects initially received 30 mg/0.3 mL of sapablursen by SC injection once every four weeks up to Week 105. After the protocol Amendment 2 the dose was increased to a maximum of 160 mg once every 4 weeks.
Arm/Group | Cohort A: Sapablursen | Cohort B: Sapablursen | Cohort C: Sapablursen
Number analyzed (Participants) | 6 | 6 | 14
percentage of participants | 0 [0.0 to 45.9] | 0 [0.0 to 45.9] | 0 [0.0 to 23.2]

3. Secondary Outcome: Percentage of Participants With a ≥1.0 Milligrams of Iron Per Grams of Dry Weight of Liver (mg Fe/g) Decrease From Baseline in Liver Iron Concentration (LIC) at Week 53
Description: Liver iron content
Time Frame: Week 53
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Sapablursen | Cohort B: Sapablursen | Cohort C: Sapablursen
Number analyzed (Participants) | 6 | 6 | 14
percentage of participants | 33.3 [4.3 to 77.7] | 50.0 [11.8 to 88.2] | 28.6 [8.4 to 58.1]

ADVERSE EVENTS:
Time Frame: From signing of informed consent to early termination (up to 733 days)
Description: Safety set included all randomized participants who received at least 1 dose of sapablursen.
Arm/Group | Cohort A: Sapablursen | Cohort B: Sapablursen | Cohort C: Sapablursen
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 1/17
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Sapablursen (N=6) | Cohort B: Sapablursen (N=6) | Cohort C: Sapablursen (N=17)
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Sapablursen (N=6) | Cohort B: Sapablursen (N=6) | Cohort C: Sapablursen (N=17)
Asthenia (General disorders) | 0 | 1 | 0
Injection Site Erythema (General disorders) | 0 | 1 | 0
Injection Site Pain (General disorders) | 1 | 0 | 0
Injection Site Pruritus (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Peripheral Swelling (General disorders) | 0 | 1 | 0
Injection Site Rash (General disorders) | 0 | 2 | 0
Vaccination Site Pain (General disorders) | 2 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 5
Fatigue (General disorders) | 4 | 1 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Adnexa Uteri Mass (Reproductive system and breast disorders) | 0 | 1 | 0
Ovulation Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 1 | 0
Blood Urine Present (Investigations) | 1 | 0 | 0
Vaccination Complication (Injury, poisoning and procedural complications) | 1 | 1 | 2
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Odontogenic Cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2
Sciatica (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Tension Headache (Nervous system disorders) | 0 | 0 | 1
Tunnel Vision (Nervous system disorders) | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Lacrimal Disorder (Eye disorders) | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal Disease (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic Mass (Hepatobiliary disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Renal Disorder (Renal and urinary disorders) | 1 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 0
Hypertonic Bladder (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Thyroid Mass (Endocrine disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0
Bacterial Vaginosis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Impetigo (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0 | 4
COVID-19 (Infections and infestations) | 3 | 0 | 11
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT04059406/Prot_SAP_001.pdf